CLINICAL TRIAL: NCT04236024
Title: The Effects of Board Game in Learning Medication Knowledge Among Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: N201912063
Record Dates: First submitted 2020-01-12; First posted 2020-01-22 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2020-12

CONDITIONS: Knowledge
Keywords: Nursing students; Board game; Medication knowledge

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The students in this group will learn medication knowledge by using board game.
  Interventions: Other: Board game
- Comparison group (Active Comparator): The students in this group will learn medication knowledge through tradition lecture.
  Interventions: Other: Traditional lecture

INTERVENTIONS:
Other: Board game — The students in the experimental group will play board game to learn medication about 30-60 minutes.
  Arms: Experimental group
Other: Traditional lecture — The students in the comparison group will receive medication lecture using PPT slides about 30-60 minutes.
  Arms: Comparison group

SUMMARY:
Background: Maintaining patient safety is one of the primary tasks of a professional nurse. Correct identification of medicine, understanding of pharmacological mechanisms and side effects are the basic academic knowledge that each nurse must possess. Therefore, it is an important duty for nursing teachers to teach students the knowledge of drugs and use them correctly in clinical practice. In this way, the safety of patients can be guaranteed and the quality of care can be improved. Board games have been used for study in different subjects, and they all have visible effects. Their competitive and entertaining qualities make learning more interesting and allow students to learn in a pleasant atmosphere. Therefore, the purpose of this study is to examine the effectiveness of using board games to teach medication knowledge to nursing students.

Methodology: This is a randomized controlled trial study. Convenience sampling will be applied in one university in Northern Taiwan.It is expected that 60-100 participants will be recruited and randomly assigned to the experimental group and comparison group by computer. The experimental group will use board game to learn medication, while the comparison group will be taught in a traditional way. The questionnaires will be conducted before the intervention, after the intervention, and one month later. The time for completing questionnaire is about 5~15 minutes. The questionnaires include demographic information, medication knowledge questionnaire, and learning satisfaction questionnaire. This study will use SPSS 22.0 software for data analysis, including frequency, percentage, mean, standard deviation, t-test, chi-square, and generalized estimation equation (GEE).

Expected results: This study will be able to understand the effects of board games in learning medication among nursing students.

ELIGIBILITY:
Inclusion Criteria:

Nursing student The student who has not yet taken a practicum course

Exclusion Criteria:

The student who had already taken a pharmacology course or is taking a pharmacology course.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Medication knowledge at 1 month | The data will be collected at baseline,immediately after the intervention, and one month after the intervention.
  This self-developed questionnaire which was validated by 5 experts will be used to understand students' medication knowledge level. The questionnaire includes 20 questions, 1 point for correct answers, 0 points for incorrect answers or not knowing, the total score is between 0 and 20 points, the higher the score represent the higher understanding of medical knowledge.

SECONDARY OUTCOMES:
Learning satisfaction questionnaire | The data will be collected immediately after the intervention.
  This self-developed questionnaire which was validated by 5 experts will be used to understand students' sanctification level regarding learning through board game or traditional lecture.The questionnaire consists of 8 questions. It is scored using the Likert scale 5 points method. 1 point is strongly disagreeable, 2 points are disagreeable. 3 points are generally agreed. 4 points are agreed. The total score is between 8-40 points, a higher score indicates that the student is more satisfied with the teaching method.

CONTACTS AND LOCATIONS:
Overall Officials: Yeu-Hui Chuang, PhD, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Every information of the participants are classified, only the result of the research can be accessed to.